## **Cover Page**

## **Study Protocol**

## Study Title: Unilateral Strength Training and Mirror Therapy for Patients with Chronic

## **Stroke. A Pilot Randomised Controlled**

**Trial** Document creation date: July 12th 2015

NCT number [not yet assigned].

Identifiers: [NCT ID not yet assigned]

Study Protocol for Unilateral Strength Training and Mirror Therapy for Patients with Chronic Stroke. A Pilot Randomised Controlled Trial (Daniel Simpson, IT Sligo)

The intervention comprised of a home-based isometric strength training programme performed under supervision by two therapists. The participant's less-affected (LA) lower limb was strapped into an ankle brace securing the ankle joint at a 100° angle (10° plantarflexion). Subjects were seated on a chair with back support, with a knee joint angle at 120°. Following a warm-up consisting of unilateral submaximal isometric contractions, the main part of the training programme consisted of 4 sets of 5 maximal effort isometric ankle dorsiflexion contractions, performed with the LA limb only, held for 5 seconds with 5 seconds rest between repetitions and 3 minutes rest between sets. The same protocol was followed 3 times per week for 4-weeks (12 sessions).

The Unilateral Strength Training only (Cross-education) group exercised without a mirror; the Experimental Group (Mirror Therapy) group observed the reflection of the LA lower limb in the mirror while training. Prompts to focus on the reflection in the mirror were given to the Mirror Strength Training group only; other verbal cues were identical for all participants of both groups.